CLINICAL TRIAL: NCT01802918
Title: A Double-Blind, Randomized, Placebo-Controlled, Single Dose Escalation First Time in Human Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK2838232 and to Evaluate the Effect of Food and Ritonavir on GSK2838232 in Healthy Subjects
Brief Title: Single Dose Escalation Study of GSK2838232 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 116787
Record Dates: First submitted 2013-02-14; First posted 2013-03-04 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: single dose; HIV; maturation inhibitor; GSK2838232; FTIH; healthy subjects
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — GSK-2838232; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Subject in this cohort will be randomized to one of the four following treatment sequences (1 treatment per visit): ABCD, BACD, BCAD, or BCDA. Where A=Placebo, B= GSK2838232 5mg, C=GSK2838232 10mg, and D=GSK2838232 20mg
  Interventions: Drug: GSK2838232; Drug: Placebo
- Cohort 2 (Experimental): Subject in this cohort will be randomized to one of the four following treatment sequences (1 treatment per visit): EGHJ, FEHJ, FGIJ, or FGHK. Where E=Placebo, F= GSK2838232 50mg, G= GSK2838232 100mg, H= GSK2838232 50mg + food, I= Placebo + food, J= GSK2838232 10mg + RTV, K= placebo + RTV.
  Interventions: Drug: GSK2838232; Drug: Placebo; Drug: Ritonavir

INTERVENTIONS:
Drug: GSK2838232 — Bottled powder with 5, 10 and 20mg unit dose strength per single dose for re-constituted oral suspension given once daily
Drug: Placebo — Visually matching GSK2838232
Drug: Ritonavir — 100mg tablets once daily for 12 days
  Arms: Cohort 2

SUMMARY:
GSK2838232 is a novel human immune virus (HIV) maturation inhibitor being developed for the treatment of chronic HIV infection. This study is the first administration of GSK2838232 in humans to establish the initial safety, tolerability, and pharmacokinetic profile following single doses of GSK2838232 and to evaluate the effect of food and ritonavir (RTV) on GSK2838232 in healthy subjects. There will be 2 cohorts in this study. In Cohort 1, approximately 8 healthy subjects will be enrolled (6 active and 2 placebo) at each dose visit. There will be four dosing sessions for each subject with subjects randomized to receive placebo in a random sequence. In Cohort 2, approximately 8 healthy subjects will be enrolled (6 active doses and 2 placebo doses at each dose visit). Cohort 2 will have four dosing sessions for each subject with subjects randomized to receive placebo in a random sequence.

ELIGIBILITY:
Inclusion Criteria

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinically significant abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Male or female between 18 and 50 years of age inclusive, at the time of signing the informed consent. A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone >40 milli international unit [MlU]/milliliter [mL] and estradiol <40 picogram [pg]/mL [<147 picomoles /liter] is confirmatory).
* Body weight >= 50 kilograms (kg) (110 pounds.) for men and >= 45 kg (99 pounds) for women and body mass index (BMI) within the range 18.5 to 31.0 kg/meter^2 (inclusive).
* A Creatinine clearance (CLcr) >80 mL/minute (min) as determined by Cockcroft-Gault equation. CLcr (mL/min) = (140 - age) x weight / (72 x serum creatinine [Scr]) (times 0.85 if female) where age is in years, weight is in kg, and Scr is in units of milligram (mg)/deciliter (dL).
* Male subjects with female partners of child-bearing potential must agree to use contraception method. This criterion must be followed from the time of the first dose of study medication until the follow up visit.
* Subject must be capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin >= 1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Screening or baseline cardiac troponin I greater than the 99 percent cutoff (>.045 nanogram [ng]/mL by the Dimension Vista cardiac troponin I [CTNI] assay).
* Screening BNP greater than the upper limit of normal
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immuno Virus antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive urine or serum human chorionic gonadotropin (hCG) test at screening or prior to dosing on Day 1.
* Lactating females.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subjects who have asthma or a history of asthma
* A history of or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* Exclusion Criteria for 24-Hour Screening Holter are: any symptomatic arrhythmia (except isolated extra systoles), sustained cardiac arrhythmias (such as atrial fibrillation or flutter, supraventricular tachycardia (>=10 consecutive beats), complete heart block), non-sustained or sustained ventricular tachycardia (defined as >= 3 consecutive ventricular ectopic beats), any conduction abnormality (including but not specific to left or right incomplete or complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], Wolff-Parkinson-White [WPW]syndrome etc.), sinus Pauses > 3 seconds, 300 or more supraventricular ectopic beats in 24 hours, and 250 or more ventricular ectopic beats in 24 hours.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination) are: Male subjects with Heart rate <45 and >100 beats per minute (bpm) and female subjects with heart rate <50 and >100 bpm, PR <120 and >220 milliseconds (msec), QRS duration <70 and >120 msec, QT interval corrected for heart rate (Fridericia's) >450 msec. (Note: A heart rate from 100 to 110 bpm can be rechecked by ECG or vitals within 30 minutes to verify eligibility).

Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization).

Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], WPW syndrome).

Sinus Pauses > 3 seconds. Any significant arrhythmia which, in the opinion of the principal investigator OR GSK medical monitor, will interfere with the safety for the individual subject.

Non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).

* Medical history of cardiac arrhythmias or cardiac disease or a family and personal history of long QT syndrome.
* Any clinically significant abnormal echocardiogram finding. Abnormal echocardiogram findings should be discussed with the Medical Monitor prior to enrolment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-02-18 (Actual); Primary Completion 2013-11-21 (Actual); Study Completion 2013-11-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) as a measure of safety and tolerability in cohort 1 | Up to 16 weeks
  AEs will be collected from the start of Study Treatment and until 5 days post last-dose (at follow up).
Number of subjects with AEs as a measure of safety and tolerability in cohort 2. | Up to 12 weeks
  AEs will be collected from the start of Study Treatment and until 5 days post last-dose (at follow up).
Absolute values and changes over time of hematology as a measure of safety and tolerability in cohort 1. | Up to 16 weeks
Absolute values and changes over time of hematology as a measure of safety and tolerability in cohort 2 | Up to 12 weeks
Absolute values and changes over time of clinical chemistry as a measure of safety and tolerability in cohort 1. | Up to 16 weeks
Absolute values and changes over time of clinical chemistry as a measure of safety and tolerability in cohort 2. | Up to 12 weeks
Absolute values and changes over time of urinalysis as a measure of safety and tolerability in cohort 1. | Up to 16 weeks
Absolute values and changes over time of urinalysis as a measure of safety and tolerability in cohort 2 | Up to 12 weeks
Absolute values and changes over time of vital signs as a measure of safety and tolerability in cohort 1 | Up to 16 weeks.
  Vital signs include blood pressure, temperature and heart rate measurement
Absolute values and changes over time of vital signs as a measure of safety and tolerability in cohort 2. | Up to 12 weeks
  Vital signs include blood pressure, temperature and heart rate measurement
Absolute values and changes over time of ECG intervals and ECG rhythm as a measure of safety and tolerability in cohort 1. | Up to 16 weeks.
Absolute values and changes over time of ECG intervals and ECG rhythm as a measure of safety and tolerability in cohort 2. | Up to 12 weeks
Real time collection and review of heart rhythm using telemetry as a measure of safety and tolerability in cohort 1. | Up to 16 weeks.
Real time collection and review of heart rhythm using telemetry as a measure of safety and tolerability in cohort 2. | Up to 12 weeks
Composite of pharmacokinetics (PK) parameters following single dose administration of GSK2838232 in cohort 1 | PK samples will be collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, and 72 hours post dose in each dosing session and at follow up visit.
  PK parameters include: area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC [0-infinity]), area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC [0-t]), maximum observed concentration (Cmax), time to maximum observed concentration (Tmax), observed concentration at 24hour post-dose (C24), last observed quantifiable concentration (Ct), lag time before observation of drug concentrations in sampled matrix (tlag), terminal half-life (t1/2), and apparent oral clearance (CL/F).
Composite of pharmacokinetics parameters following single dose administration of GSK2838232 in cohort 2. | PK samples will be collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, and 72 hours post dose in each dosing session and at follow up visit.
  PK parameters include: AUC (0-infinity), AUC (0-t), Cmax, Tmax, C24, Ct, tlag, t1/2 and CL/F.

SECONDARY OUTCOMES:
Composite of pharmacokinetics parameters following single dose administration of GSK2838232 with and without food in cohort 2. | PK samples will be collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, and 72 hours post dose in each dosing session and at follow up visit.
  PK parameters include: AUC (0-infinity), AUC (0-t), Cmax, Tmax, C24 and t1/2. Food will be normal fat meal.
Composite of pharmacokinetics parameters following single dose administration of GSK2838232 with co-administration of ritonavir in cohort 2. | PK samples will be collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, and 72 hours post dose in each dosing session and at follow up visit.
  PK parameters include: AUC (0-infinity), AUC (0-t), Cmax, Tmax, C24 and t1/2.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

REFERENCES:
- See also: Results for study 116787 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116787?search=study&search_terms=116787#rs